CLINICAL TRIAL: NCT02709876
Title: Autologous Bone Marrow-Derived CD34+, CD133+, and CD271+ Stem Cell Transplantation for Retinitis Pigmentosa
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-RP1
Record Dates: First submitted 2016-02-26; First posted 2016-03-16 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cells (Experimental): Intravitreal Injection of bone marrow derived CD34+, CD133+, CD271+ stem cells.
  Interventions: Biological: Stem Cell Transplantation

INTERVENTIONS:
Biological: Stem Cell Transplantation — Bone marrow-derived CD34+, CD133+, CD271+ stem cells in 1.0 ml normal saline will be injected into the vitreous cavity.

SUMMARY:
A single arm, single center trial to evaluate the safety and efficacy of autologous purified populations of bone-marrow derived stem cells in patients with Retinitis Pigmentosa (BM-SCs) through a 48 month follow up period.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is an inherited disorder of the photoreceptor cells in the retina. Patients may lose vision since they were young or later in life. Currently, there are more than 60 genes identified as the cause of this condition, one of which, RPE65, has been studied in several gene therapy trials for Leber congenital amaurosis with promising results. Another treatment approach for RP is stem cell therapy. Studies in animal models of RP have shown that subretinal injection of bone marrow-derived mesenchymal stem cells may delay degenerative changes of photoreceptor cells. This is a single arm, single center trial to assess the safety and efficacy of purified adult autologous bone marrow derived CD34+, CD133+, and CD271+ stem cells through a 48 month follow-up period. The combination of these three cell types was based on their diverse potentialities to differentiate into specific functional cell types to regenerate damaged retinal tissue, and the availability of clinical-grade purification system (CliniMACS) and microbeads to purify the target cell populations in clinically-approved methods.

ELIGIBILITY:
Inclusion Criteria:

* Retinitis pigmentosa patients diagnosed by ophthalmologists
* Visual acuity (measured with ETDRS) less than or equal to 20/70 and visual field below 30° central in both eyes.
* Best corrected visual acuity less than 6/120 by Snellen visual acuity chart

Exclusion Criteria:

* Other eye conditions that could mask the interpretation of the results
* Unable to return for follow up
* Underlying diseases including asthma, heart failure, myocardial infarction, liver failure, renal failure
* Pregnant and lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
ETDRS Visual acuity change | 12 months from baseline

SECONDARY OUTCOMES:
Quality of Life: Questionnaire VFQ-25 (Visual Function Questionnaire-25) | 12 months from baseline
Color Vision: Ishihara Color Test | 12 months from baseline
Contrast sensitivity: CSV-1000E | 12 months from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Stem Cells Arabia, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes